CLINICAL TRIAL: NCT07315646
Title: The PAINLESS Study: Pain Associated wIth traditioNal Versus uLtrasound guidEd iuS (Intra Uterine System) inSertion
Brief Title: Pain Associated wIth traditioNal Versus uLtrasound guidEd iuS (Intra Uterine System) inSertion
Acronym: PAINLESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Imelda Hospital, Bonheiden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONZ-2025-0220
Record Dates: First submitted 2025-12-08; First posted 2026-01-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Intra-uterine Device Placement
Keywords: intra-uterine device placement; TAS-technique; contraception use; uterine bleeding heavy; menopausal bleeding; family planning
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The TAS (transabominal ultrasound) insertion technique (Experimental): This new technique uses transabdominal sonography during IUS placement. The placement under constant visualization eliminates the need for Pozzi tenaculum and uterine soundings.
  Interventions: Procedure: IUS (intrauterine system) insertion
- The Traditional Technique (Active Comparator): The traditional technique for an IUS insertion uses a speculum after which a Pozzi tenaculum is placed on the cervix so that the uterus is brought into the stretching position by means of traction. The cavum is then measured by a uterine sound. These actions and the use of these instruments can contribute to the pain experience during insertion.
  Interventions: Procedure: IUS (intrauterine system) insertion

INTERVENTIONS:
Procedure: IUS (intrauterine system) insertion — Intra-uterine device insertion (technique based on randomization arm)

SUMMARY:
Rationale: The 2019 Belgian Health Survey shows that the combined oral contraceptive pill is the most commonly used form of contraception. However, the Pearl index of Long-acting reversible contraceptive (LARC) methods is significantly better (perfect and typical use <0.5) compared to the combined oral contraceptive pill (perfect use <1.0, typical use 2-9). An IUS is an example of a LARC method. IUS insertion might be painful. Because of this, women may be reluctant to opt for an IUS. The traditional technique for an IUS insertion uses a speculum after which a Pozzi tenaculum is placed on the cervix so that the uterus is brought into the stretching position by means of traction. The cavum is then measured by a uterine sound. These actions and the use of these instruments can contribute to the pain experience during insertion. The new technique, transabdominal sonographic (TAS) insertion, could reduce the pain experience during insertion. This new technique uses transabdominal sonography during IUS placement. The placement under constant visualization eliminates the need for Pozzi tenaculum and uterine soundings. Little high quality studies have been conducted on the advantages and disadvantages of the TAS technique as demonstrated by a non-published systematic review of the literature.

Research question/goal: Is the insertion of an IUS (Kyleena/Mirena) using the TAS technique less painful than the traditional technique?

Study design: A randomized trial (RCT) in which the subject is blinded to the insertion technique.

Study population: Women wishing an IUS (Kyleena & Mirena)

Primary and secondary outcomes:

The primary outcomes are the pain during insertion (Numeric Rating Scale (NRS) score 0-10) and dislocation: non-fundal position (> 3mm fundal distance postinsertion) in the uterine cavity (Y/N).

Secondary outcomes include the average and worst pain in the first week after insertion (NRS 0-10), expulsion of the IUS, perforation of the uterine wall, failure of insertion, the occurrence of vagal symptoms, use of pain relief the first 7 days after placement, subject satisfaction about the procedure, successful IUS placement.

ELIGIBILITY:
Inclusion Criteria:

* Women between18 years and 60 years (at the time of signing the ICF)
* Who wish to have an IUS (Kyleena/Mirena) for reasons of family planning, conservative treatment for abnormal uterine bleeding or as part of hormonal treatment for menopausal symptoms
* Dutch-speaking subjects

Exclusion Criteria:

* History of difficult IUS placement
* Known cervical stenosis
* Asherman's syndrome
* Standard contraindications to an IUS (eg breast cancer, recent deep vein thrombosis, anatomical uterine abnormalities, pregnancy, acute PID, cervicitis, vaginitis or any lower genital tract infection, cervical or endometrial malignancy, history of septic abortion or postpartum endometritis in the last 3 months,.. )
* Current pelvic inflammatory disease
* Pregnancy
* Trophoblastic disease
* Known cervical or endometrial carcinoma
* Patients who have the profession of midwife, nurse or doctor.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain during insertion of the IUS | From enrollment to the intervention date (IUS placement)
  Pain during insertion, reported by the subject on a Numeric Rating Scale (NRS scale) 0-10
Dislocation | From enrollment to intervention date (IUS placement)
  Dislocation: non-fundal position (> 3mm fundal distance postinsertion) in the uterine cavity (Y/N)

SECONDARY OUTCOMES:
Expulsion | During of directly after the intervention (IUS placement)
  Expulsion of the IUS during the procedure (Y/N)
Failure of insertion | During the procedure of IUS placement
  Failure of insertion (yes/no)
vagal symptoms | During IUD insertion
  Vagal symptoms: paillor, sweating, syncope (yes/no)
Pain experience during 7 days after placement | During the 7 days after IUS insertion
  Pain experience (average and worst pain) during 7 days after placement (NRS 0-10)
Pain relief taken during the 7 days after IUS placement | During the 7 days after IUS placement
  Pain relief taken during the 7 days after placement (Y/N, if yes specify in text field (what, dose, timing))
Satisfaction with the procedure | Seven days after IUS placement
  Subject satisfaction with the technique (5 point Likert scale)
Successful IUS placement | Directly after IUS insertion procedure
  Successful IUS placement (Y/N)
Perforation | During IUS placement
  Perforation: IUS perforates the uterine wall (Y/N). Characterized by sharp pain and blood loss during insertion, ultrasound extrauterine position in total perforation or positioned in the myometrium in partial perforation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Weyers, MD, PhD, Principal Investigator — University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No